CLINICAL TRIAL: NCT06866366
Title: Impact of the Use of Resource® Diabet Plus on Metabolic Control in Patients With T2DM Who Are Malnourished or at Risk of Malnutrition
Brief Title: Retrospective, Multicenter, Single-arm, Observational Study, With Data From Patients With T2DM With Malnutrition or at Risk, Who Were Prescribed Resource® Diabet Plus as a Hypercaloric and Hyperproteic Specific Formula for Patients With T2DM
Acronym: ReDiPLUS
Status: Completed | Type: Observational
Sponsor: Outcomes'10 (Network)
Collaborators: Nestlé Health Science Spain (Industry)
Responsible Party: Sponsor
Other Study IDs: NES-2023-152-RET-DP
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Malnourished Elderly; Malnourishment; Diabetes Mellitus Type 2
Keywords: DRM; Disease - realted malnutrition; Diabetes-specific formula; Metabolic control; Oral nutritional supplementation; DSF; T2D
MeSH Terms: conditions — Malnutrition; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with T2DM with malnutrition or at risk, who were prescribed: Resource® Diabet Plus

SUMMARY:
This retrospective multicentre study aims to provide real-world evidence of the effectiveness of Resource® Diabet Plus as supplementation tool for T2DM patients with malnutrition or at risk of malnutrition, under conditions of routine clinical practice in Spain.

DETAILED DESCRIPTION:
Disease-related malnutrition (DRM) is a nutritional imbalance caused by a nutrient deficiency resulting from one or more underlying pathologies. It is the main cause of malnutrition in developed countries, with a prevalence of around 30 million people in Europe in 2020. In Spain, it is estimated that around 20-50% of hospitalized patients suffer from DRM, both in acute and chronic conditions. One of the chronic diseases where malnutrition is associated with higher mortality and increased hospital admissions is Type 2 Diabetes Mellitus (T2DM), particularly in the elderly. T2DM is currently one of the most prevalent chronic diseases worldwide, affecting about 10% of the adult population in 2021. Approximately 90% of diagnosed cases of diabetes are type 2, which is not autoimmune-mediated, unlike type 1 (T1DM). T2DM typically develops over time due to factors such as obesity, sedentary lifestyle, high-calorie diets, and aging. Additionally, malnutrition risk is increased in patients with T2DM, which leads to a poorer prognosis.

For the treatment of DRM in diabetic patients, as in other chronic conditions, clinical guidelines recommend a personalized nutritional plan tailored to the patient's needs and characteristics, primarily focused on increasing dietary calorie intake. If this is insufficient, oral nutritional supplements may be necessary. From a clinical perspective, oral nutritional supplements address malnutrition while offering clinical and functional benefits. In diabetic and malnourished patients, it is crucial to maintain good metabolic and glycemic control, which requires diabetes-specific formulas (DSFs).

Unlike standard formulas, which are typically high in carbohydrates, low in lipids, and lack dietary fiber, DSFs contain carbohydrates with low glycemic indices and also include fiber. The purpose of these formulas is to improve the nutritional status of patients without negatively affecting their glycemic profile, aiming for adequate glycated hemoglobin (HbA1c) levels - values under 7% are generally recommended for this population.

Prospective observational studies in malnourished T2DM patients have shown that supplementation with a DSF for at least 12 weeks improves patients' functional and nutritional status, enhances biochemical markers, and does not increase postprandial glucose levels. Additionally, the use of these formulas benefits glycemic and metabolic control in the short and medium term, potentially improving diabetes management and its associated comorbidities, while reducing long-term complications and mortality.

A retrospective study conducted in 2015 in the Spanish diabetic population suggested that this type of DSF may reduce HbA1c in the medium term, facilitating glycemic control and reducing the negative effects of glycemic fluctuations. This could result in a reduced need for insulin as an antidiabetic treatment.

The existing evidence supports the benefits of DSFs in diabetic patients by helping to maintain metabolic control and improving nutritional, functional, and clinical outcomes. These improvements are associated with fewer hospital visits and admissions. However, more studies are needed to confirm the advantages of using these nutritional formulas specifically designed for diabetic and malnourished patients. Although they are somewhat more expensive than standard supplements, they help patients achieve better metabolic control, which can ultimately lead to lower healthcare costs.

Few retrospective studies have been conducted in the field of nutrition for diabetic and malnourished patients. Most available data come from prospective studies or literature reviews. However, the nature of retrospective real-world studies allows for the assessment of DSF use in a specific population over a relatively short time period, reflecting how malnourished diabetic patients are managed in clinical practice.

This retrospective study aims to provide real-world evidence on the effectiveness of Resource® Diabet Plus supplementation as a DSF in diabetic patients with malnutrition or at risk, under routine clinical practice conditions in Spain.

OBJECTIVES OF THE STUDY

Primary Objective:

- To assess the effects of Resource® Diabet Plus on glycemic control in patients with T2DM who are malnourished or at risk, 12 and 24 weeks after initiation of nutritional therapy.

Secondary Objectives:

* To assess the effects of Resource® Diabet Plus on metabolic control in malnourished or at-risk T2DM patients at 12 and 24 weeks after treatment initiation.
* To describe the evolution of nutritional and functional status in T2DM patients who are malnourished or at risk, 12 and 24 weeks after starting Resource® Diabet Plus.
* To describe the presence of gastrointestinal symptoms in patients treated with Resource® Diabet Plus.
* To analyze healthcare resource utilization and associated costs after 24 weeks of treatment with Resource® Diabet Plus.

METHODOLOGY

Study Design and Scope:

This is a retrospective, multicenter, single-arm observational study including data from patients at risk of malnutrition identified through validated screening tools or with DRM diagnosed using GLIM criteria, who were prescribed a specific hypercaloric and high-protein formula for diabetic patients: Resource® Diabet Plus. The study will be conducted in the Endocrinology and Nutrition Departments of four Spanish hospitals.

Resource® Diabet Plus must have been prescribed between two years and 24 weeks prior to the study start date. Clinical history data will be collected at the time of prescription (index date, V0), and follow-up data will be collected at 12 weeks (V1) and 24 weeks (V2), allowing a two-week window to adapt to each center's clinical practice. Investigators will have a 3-month window for patient identification and data collection.

Study Product: Resource® Diabet Plus

The study product, Resource® Diabet Plus, is a high-protein and hypercaloric (1.6 kcal/mL) oral nutritional formula with fiber, made from milk protein and 100% soluble fiber. It is suitable for patients with type 1 diabetes, T2DM, or hyperglycemia with increased energy and protein requirements and conditions involving nutritional risk or malnutrition.

Resource® Diabet Plus is presented in 200 mL bottles, each containing:

* 18 g of protein
* 5 g of soluble fiber
* 7.2 g of monounsaturated fatty acids from vegetable oils

Additionally, Resource® Diabet Plus contains slowly absorbed carbohydrates with a glycemic index below 55, making it appropriate for achieving metabolic targets while maintaining glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years.
* Outpatients or hospitalised patients, at discharge with a diagnosis of type 2 Diabetes.
* Patients at risk of malnutrition detected by validated screening tools or with DRM diagnosed by GLIM criteria.
* Patients who have been prescribed 1-2 bottles/day of Resource® Diabet Plus following the conditions of use of its technical data sheet, in the last 2 years, with at least 24 weeks of evolution recorded in the clinical history.
* Patients who have Hb1Ac data in the medical record on the index date and during evolution.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Patients who required any other type of nutritional supplementation during the study period (parenteral/enteral).
* Patients with severe renal insufficiency (glomerular filtration rate < 30mL/min/1.73m2) at the time of selection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic patient with malnutrition or at risk of malnutrition, treated for it in hospitals of the national network who have been prescribed 1-2 bottles/day of Resource® Diabet Plus
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-07-13 (Actual); Study Completion 2025-07-13 (Actual)

PRIMARY OUTCOMES:
Glycaemic control | In 12 and 24 weeks from baseline visit
  Changes in HbA1c, meaning a percentage less than 7, good glycaemic control.

SECONDARY OUTCOMES:
Metabolic control | In 12 and 24 weeks from baseline visit
  Changes in total cholesterol, HDL, LDL and triglycerides. Calculating the number and percentage of patients who increase, decrease or maintain them and those who achieve good metabolic control (defined as: total cholesterol<185mg/dL, HDL>40mg/dL, LDL<100mg/dL and triglycerides<150mg/dL).
Nutritional and functional status | In 12 and 24 weeks from baseline visit
  Changes in GLIM criteria, arm circumference, calf circumference and prehensile strength
Gastrointestinal tolerance | In 12 and 24 weeks from baseline visit
  By monitoring gastrointestinal symptomatology
Healthcare resource use and associated costs | During 24 weeks from baseline visit
  Data will be collected on hospitalisations, emergency department visits and specialist visits (all of which are related to malnutrition) for patients during the 24 weeks of treatment. Changes in the patient's anti-diabetic medication, if any, will also be collected. The cost will be calculated by extrapolating each resource to the cost as listed in eSalud and BOT PLUS

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: No